CLINICAL TRIAL: NCT04945967
Title: A New Intervention Method to Enhance Oral Feeding Ability in Premature Infants: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Luh Karunia Wahyuni, Sp.KFR(K), M.D., Pediatric Physiatrist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-03-0235
Record Dates: First submitted 2021-05-28; First posted 2021-06-30 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Feeding; Difficult, Newborn; Premature
Keywords: Premature Infant; Oral Feeding Ability; Therapeutic Positioning; Oromotor Intervention
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Premature infants at 28 to 34 weeks of gestational age and has achieved oral feeding readiness but unable to achieve safe and efficient oral feeding will be divided into 2 groups for intervention: New method and conventional method interventions.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Method (Experimental): This intervention will be given once a day, 30 minutes before feeding schedule based on the neonatologist. Each session of intervention will take time about 18 minutes.
  Interventions: Procedure: New Method
- Conventional Method (Active Comparator): This intervention will be given once a day, 30 minutes before feeding schedule based on the neonatologist. Each session of intervention will take time about 15 minutes.
  Interventions: Procedure: Conventional Method

INTERVENTIONS:
Procedure: New Method — Physiological flexion in therapeutic positioning, oral stimulation, stimulation of synergistic movements, and stimulation for non-nutritive sucking by using special designed pacifier for premature infant.
  Arms: New Method
Procedure: Conventional Method — Oral stimulation and non-nutritive sucking stimulation using usual pacifier.
  Arms: Conventional Method

SUMMARY:
Indonesia is the fifth country with the highest number of premature infants in the world. Research has shown that as many as 40% to 70% of premature infants exhibit both immature and atypical feeding skills and those requiring respiratory support and those experiencing delays in beginning oral feeding are most often affected.

Majority of premature infants have poorly developed suck and swallow mechanisms. The neurological immaturity, abnormal muscle tone, depressed oral reflexes, and difficulty in regulating state, can decrease the quality of infant's oral motor skills and the quantity of intake. For these reasons many high-risk infants are unable to tolerate oral feeding from birth and have difficulty making the transition from tube feedings to functional oral feeding. This transition to full oral feeding is an important competency for the infant to attain prior to discharge home. Delays in discharge are often secondary to feeding difficulties, leading to increased medical costs.

Currently a number of treatment strategies exist to facilitate oral feeding in premature infants. These include environmental/physical modifications such as eliminating external stimuli during feedings, using therapeutic nipples to manipulate flow rate, positioning and swaddling to support the motor system and improve flexion, and oral motor intervention including Non-nutritive sucking (NNS) stimulation and oral/perioral stimulation. There are known various methods of oral and perioral stimulations. Recent study claimed that oral stimulations combined with non-nutritive sucking stimulation in premature infants for at least 10 days period could facilitate oral feeding ability.

The therapy of new method intervention that will be studied in this research was a combination of physiological flexion in therapeutic positioning with specific swaddling techniques, oral stimulation, stimulation of synergistic movements, and stimulation of non-nutritive sucking using a special designed pacifier according to the size of premature infant's oral cavity.

The objective of this study is to determine the time span required for premature infant to achieve safe and efficient oral feeding after new method intervention. Therefore, this new method expectedly can be used as an intervention to improve oral feeding ability in premature infant.

DETAILED DESCRIPTION:
This study was designed as a double-blinded and randomized controlled trial, which was held from August 2021 until November 2021 in five tertiary hospitals in Jakarta area: Dr. Cipto Mangunkusumo National Central General Hospital, Harapan Kita Women & Children's Hospital, Bunda Women & Children's Hospital, Pasar Rebo Regional General Hospital, and Budi Kemuliaan General Hospital. Premature infants born in 28-34 weeks who has achieved oral feeding readiness but had not achieved oral feeding ability will be recruited as participants. Subjects were then randomized and assigned to New method and Conventional method intervention groups. The total number of sample size was 70 subjects.

Both interventions were given once a day, 30 minutes before the infant's feeding schedule. After each session of intervention was done, participant will be evaluated for oral feeding ability.

Participant will be in semi-upright position, using peristaltic plus for low-birth-weight pacifier in SS size. The volume of fluids feed will be decided based on neonatologist's assessment. Participant was stated to achieve oral feeding ability if participant was able to swallow more than 30% of the volume set by the neonatologist for the first 5 minutes at a rate of more than or equal to 1.5 ml / minute and without signs of aspiration. If the results of the evaluation show that the participant has not been able to achieve safe and efficient oral feeding, intervention will be terminated. If the participant has not fulfilled the criteria, intervention will be continued. However, if the participant became unstable after given each intervention, then intervention will be halted and will be repeated again in the next feeding schedule. After 3 consecutive trials and the participant is still unstable while given intervention, then the participant will be put in drop out category.

Statistical analysis will be conducted using SPSS ver. 20.0. The level of significance was set at <0.05. Interim analysis will be conducted in this research and will be done in three steps:

1. Basic data analysis for comparing distribution between two intervention groups with descriptive analysis.
2. Bivariate analysis using chi-square.
3. Multivariate analysis using logistic regression if there are incomparable basic data variables.

ELIGIBILITY:
Inclusion Criteria:

1. Premature infants born 28 to 34 weeks of gestational age
2. Has achieved oral feeding readiness in the form of :

   * Stable cardiorespiratory status
   * Fully feed through orogastric tube of 120ml/kg/day without vomiting or bloating
   * Strong and rhythmic non-nutritive sucking (NNS), measured objectively using sucking mechanism evaluation system (5 to 10 non-nutritive sucks per burst, the repetitive pattern was stable, with a pause of 4 to 9 seconds, and the amplitude was -16.7 to -87 mmHg)
3. Parent/guardian give consent to participate

Exclusion Criteria:

1. Craniomaxillofacial malformation
2. Neonatal asphyxia with 5-minute APGAR score is less than 7
3. Grade 3 and 4 intraventricular hemorrhage
4. Using endotracheal tube at the time of assessment

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Time Span to Achieve Safe and Efficient Oral Feeding After New Method Intervention | 1st day after the first session of New method intervention to oral feeding ability achievement
  Time span is measured in days. New method intervention will be given once a day. After New method intervention is done, participant will be evaluated for safe and efficient oral feeding. If the participant has already fulfilled the criteria in safe and efficient oral feeding, intervention will be ended. If participant has not fulfilled the criteria, intervention will be continued.
Time Span to Achieve Safe and Efficient Oral Feeding After Conventional Method Intervention | 1st day after the first session of conventional method intervention to oral feeding ability achievement
  Time span is measured in days. Conventional method intervention will be given once a day. After conventional method intervention is done, participant will be evaluated for safe and efficient oral feeding. If the participant has already fulfilled the criteria in safe and efficient oral feeding, intervention will be ended. If participant has not fulfilled the criteria, intervention will be continued.

CONTACTS AND LOCATIONS:
Overall Officials: Luh K. Wahyuni, MD, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (1):
- Dr. Cipto Mangunkusumo National General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No